CLINICAL TRIAL: NCT03979638
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover, Dose Escalation Study of BLU-5937 in Subjects With Unexplained or Refractory Chronic Cough (RELIEF)
Brief Title: A Dose Escalation Study of BLU-5937 in Unexplained or Refractory Chronic Cough
Acronym: RELIEF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was terminated due to the impact of the COVID-19 on trial activities. 68 patients with refractory chronic cough were enrolled with 52 completing treatment
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUS-P2-01; 2019-000375-16 (EudraCT Number)
Record Dates: First submitted 2019-06-06; First posted 2019-06-07 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2020-04

CONDITIONS: Chronic Refractory Cough
Keywords: Unexplained or refractory chronic cough, P2X3 antagonists
MeSH Terms: conditions — Chronic Cough | interventions — BLU-5937

STUDY DESIGN:
Intervention Model Description: Two-arm, Two-Period, crossover assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BLU-5937 oral tablet BID (Experimental): Randomized crossover design of 4 different doses (25, 50, 100, 200 mg BID) of BLU-5937 tablets to be administered orally BID
  Interventions: Drug: BLU-5937
- Placebo oral tablet BID (Placebo Comparator): Randomized crossover design of matching placebo tablets to be administered orally BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BLU-5937 — Four escalating doses of BLU-5937 administered BID over the course of the study
  Arms: BLU-5937 oral tablet BID
Drug: Placebo — Matching placebo for BLU-5937
  Arms: Placebo oral tablet BID

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, crossover, dose escalation study of BLU-5937 in subjects with unexplained or refractory chronic cough

DETAILED DESCRIPTION:
This study will have two 16-day treatment periods (four escalating doses or matching placebo at four days interval) separated by a 10 to 14-day washout period. There will be a 14-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained or refractory chronic cough for at least one year
* Chest radiograph or CT thorax within the last 60 months not demonstrating any abnormality considered to be significantly contributing to the chronic cough
* Cough count of ≥ 10 per hour (Awake Cough Count) at Screening
* Score of ≥ 40mm on the Cough Severity VAS at Screening
* Women of child-bearing potential must have a negative serum pregnancy test at Screening
* Women of child-bearing potential must use a highly effective contraception method from Screening through the Follow-Up Visit
* Male subjects and their partners of child-bearing potential must use 2 methods of acceptable birth control

Exclusion Criteria:

* Current smoker or individuals who have given up smoking within the past 6 months, or those with >20 pack-year smoking history
* Diagnosis of COPD, bronchiectasis, idiopathic pulmonary fibrosis
* Treatment with an ACE-inhibitor as the potential cause of a subject's cough, or requiring treatment with an ACE-inhibitor during the study, or within 12 weeks prior to the Screening Visit
* FEV1/FVC < 60%
* History of upper respiratory tract infection or recent significant change in pulmonary status within 4 weeks of the Baseline Visit
* History of concurrent malignancy or recurrence of malignancy within 2 years prior to Screening
* History of a diagnosis of drug or alcohol dependency or abuse within the last 3 years
* Clinically significant abnormal electrocardiogram (ECG) or laboratory tests at Screening
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacky Smith, MD, Ph.D., Principal Investigator — University of Manchester
Locations (16):
- United States (8):
  - Allergy Associates Medical Group Inc., San Diego, California
  - Allergy & Asthma Associates of Santa Clara Valley, San Jose, California
  - Centre for Cough, Largo, Florida
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - National Allergy & Asthma Research, Charleston, South Carolina
  - Diagnostics Research Group, San Antonio, Texas
  - Allergy Asthma & Sinus Center, Greenfield, Wisconsin
- United Kingdom (8):
  - Belfast City Hospital, Belfast
  - Castle Hill Hospital, Cottingham
  - University Hospitals of Leicester, Leicester
  - Prince Phillip Hospital, Llanelli
  - King's College Hospital, London
  - Royal Brompton Hospital, London
  - Manchester Clinical Research Facility, Manchester
  - North Tyneside General Hospital, North Shields

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 16 clinical trial sites in the United-Kingdom and in United States.
Pre-assignment Details: A total of 68 participants were randomized to receive the study drug (BLU-5937) followed by placebo (33 participants) or placebo followed by the study drug (35 participants).
Groups:
- BLU-5937 > Placebo: Randomized crossover design of 4 different doses (25, 50, 100, 200 mg BID) of BLU-5937 tablets to be administered orally BID
  BLU-5937: Four escalating doses of BLU-5937 administered BID over the course of the study followed by matching Placebo
- Placebo > BLU-5937: Randomized crossover design of matching placebo tablets to be administered orally BID
  Placebo: Matching placebo for BLU-5937 follow by four escalating doses of BLU-5937
Period: Period 1
Arm/Group | BLU-5937 > Placebo | Placebo > BLU-5937
Started | 33 | 35
Completed | 26 | 28
Not Completed | 7 | 7
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Study terminated by Sponsor | 1 | 3
Not completed — Protocol Violation | 1 | 0
Period: Period 2
Arm/Group | BLU-5937 > Placebo | Placebo > BLU-5937
Started | 26 | 28
Completed | 25 | 27
Not Completed | 1 | 1
Not completed — Study terminated by Sponsor | 1 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all randomized participants who have received at least 1 dose of study drug.
Groups:
- Placebo > BLU-5937: Randomized crossover design of matching placebo tablets to be administered orally BID
  Placebo: Matching placebo for BLU-5937 followed by four escalating doses of BLU-5937
- Total: Total of all reporting groups
Arm/Group | BLU-5937 > Placebo | Placebo > BLU-5937 | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (11.49) | 63.7 (9.70) | 64.0 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 29 | 34 | 63
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 33 | 33 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Awake Objective Cough Frequency on Log-transformed Scale
Description: Change in awake cough frequency (average hourly cough frequency while the subject is awake ) evaluated using the VitaloJAK cough monitor with 24-hour sound recordings collected
Time Frame: Period 1: baseline (Day 0) and 24 hours after Day 4, 8, 12, 16 doses ; Period 2: baseline (Day 30) and 24 hours after Day 34, 38, 42, 46 doses
Population: Analysis population consisted of all randomized subjects who took at least one dose of study drug and provided at least one baseline and at least one post-baseline cough frequency measurement
Measure: Least Squares Mean (95% Confidence Interval); unit: Log coughs/hour
Groups:
- BLU-5937 - 25 mg: BLU-5937 25 mg tablet administered orally BID for 4 days
- Placebo Comparator - 25 mg; Placebo Comparator - 50 mg; Placebo Comparator - 100 mg; Placebo Comparator - 200 mg: Matching Placebo for BLU-5937 administered orally BID for 4 days
- BLU-5937 - 50 mg: BLU-5937 50 mg tablet administered orally BID for 4 days
- BLU-5937 - 100 mg: BLU-5937 100 mg tablet administered orally BID for 4 days
- BLU-5937 - 200 mg: BLU-5937 200 mg tablet administered orally BID for 4 days
Arm/Group | BLU-5937 - 25 mg | Placebo Comparator - 25 mg | BLU-5937 - 50 mg | Placebo Comparator - 50 mg | BLU-5937 - 100 mg | Placebo Comparator - 100 mg | BLU-5937 - 200 mg | Placebo Comparator - 200 mg
Number analyzed (Participants) | 60 | 59 | 59 | 58 | 56 | 58 | 58 | 58
Log coughs/hour | -0.19 [-0.29 to -0.08] | -0.07 [-0.19 to 0.05] | -0.20 [-0.32 to -0.08] | -0.14 [-0.26 to -0.01] | -0.25 [-0.40 to -0.09] | -0.17 [-0.30 to -0.04] | -0.33 [-0.49 to -0.17] | -0.14 [-0.29 to 0.00]
Statistical Analysis 1: Comparison: BLU-5937 - 25 mg vs Placebo Comparator - 25 mg; Test type: Superiority; p = 0.1424, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -10.8, 95% CI 2-sided [-23.5 to 4.0] — Percent change difference between BLU-5937 and placebo was estimated by 100 x [e^diff - 1] where 'e' = exponent of difference; and 'diff' = the treatment mean difference from mixed model of change from baseline based on log-transformed data
Statistical Analysis 2: Comparison: BLU-5937 - 50 mg vs Placebo Comparator - 50 mg; Test type: Superiority; p = 0.4602, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -6.1, 95% CI 2-sided [-20.8 to 11.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: BLU-5937 - 100 mg vs Placebo Comparator - 100 mg; Test type: Superiority; p = 0.4181, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -7.8, 95% CI 2-sided [-24.4 to 12.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: BLU-5937 - 200 mg vs Placebo Comparator - 200 mg; Test type: Superiority; p = 0.0855, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -16.7, 95% CI 2-sided [-32.3 to 2.6] — [estimate comment as in outcome 1, analysis 1]

2. Other Pre Specified Outcome: Change in Awake Cough Frequency on Log-transformed Scale in the Subgroup of Participants With Awake Cough Frequency > or = 20 Coughs/Hour at Baseline
Description: Change in awake cough frequency (average hourly cough frequency while the subject is awake) in the a pre-specified subgroup of participants with awake cough frequency > or = 20 coughs/hour at baseline evaluated using the VitaloJAK cough monitor with 24-hour sound recordings collected
Time Frame: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Log coughs/hour
Arm/Group | BLU-5937 - 25 mg | Placebo Comparator - 25 mg | BLU-5937 - 50 mg | Placebo Comparator - 50 mg | BLU-5937 - 100 mg | Placebo Comparator - 100 mg | BLU-5937 - 200 mg | Placebo Comparator - 200 mg
Number analyzed (Participants) | 46 | 46 | 45 | 46 | 44 | 47 | 45 | 46
Log coughs/hour | -0.23 [-0.34 to -0.11] | 0.00 [-0.09 to 0.10] | -0.29 [-0.42 to -0.15] | -0.09 [-0.21 to 0.03] | -0.33 [-0.51 to -0.16] | -0.12 [-0.25 to 0.01] | -0.41 [-0.58 to -0.24] | -0.09 [-0.23 to 0.05]
Statistical Analysis 1: Comparison: BLU-5937 - 25 mg vs Placebo Comparator - 25 mg; Test type: Superiority; p = 0.0010, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -20.3, 95% CI 2-sided [-29.9 to -9.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BLU-5937 - 50 mg vs Placebo Comparator - 50 mg; Test type: Superiority; p = 0.0186, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -17.7, 95% CI 2-sided [-29.9 to -3.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: BLU-5937 - 100 mg vs Placebo Comparator - 100 mg; Test type: Superiority; p = 0.0320, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -19.4, 95% CI 2-sided [-33.9 to -1.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: BLU-5937 - 200 mg vs Placebo Comparator - 200 mg; Test type: Superiority; p = 0.0026, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -27.0, 95% CI 2-sided [-40.3 to -10.8] — [estimate comment as in outcome 1, analysis 1]

3. Other Pre Specified Outcome: Change in Awake Cough Frequency on Log-transformed Scale in the Subgroup of Participants With Awake Cough Frequency > or = Median (32.4 Coughs/Hour) at Baseline
Description: Change in awake cough frequency (average hourly cough frequency while the subject is awake) in the a pre-specified subgroup of participants with awake cough frequency > or = median (32.4 coughs/hour) at baseline evaluated using the VitaloJAK cough monitor with 24-hour sound recordings collected
Time Frame: Period 1: baseline (Day 0) and 24 hours after Day 4, 8, 12,16 doses ; Period 2: baseline (Day 30) and 24 hours after Day 34, 38, 42, 46 doses
Measure: Least Squares Mean (95% Confidence Interval); unit: Log coughs/hour
Arm/Group | BLU-5937 - 25 mg | Placebo Comparator - 25 mg | BLU-5937 - 50 mg | Placebo Comparator - 50 mg | BLU-5937 - 100 mg | Placebo Comparator - 100 mg | BLU-5937 - 200 mg | Placebo Comparator - 200 mg
Number analyzed (Participants) | 28 | 30 | 28 | 31 | 27 | 31 | 28 | 31
Log coughs/hour | -0.31 [-0.45 to -0.18] | 0.02 [-0.11 to 0.15] | -0.42 [-0.55 to -0.28] | -0.08 [-0.22 to 0.05] | -0.44 [-0.60 to -0.27] | -0.09 [-0.24 to 0.06] | -0.49 [-0.68 to -0.31] | -0.10 [-0.24 to 0.03]
Statistical Analysis 1: Comparison: BLU-5937 - 25 mg vs Placebo Comparator - 25 mg; Test type: Superiority; p = 0.0005, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -28.1, 95% CI 2-sided [-39.5 to -14.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BLU-5937 - 50 mg vs Placebo Comparator - 50 mg; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -28.4, 95% CI 2-sided [-39.7 to -15.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: BLU-5937 - 100 mg vs Placebo Comparator - 100 mg; Test type: Superiority; p = 0.0014, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -29.5, 95% CI 2-sided [-42.7 to -13.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: BLU-5937 - 200 mg vs Placebo Comparator - 200 mg; Test type: Superiority; p = 0.0006, Mixed Models Analysis; Intention To Treat (ITT), statistical analysis follows a Mixed Model which uses log-transformation; Estimated percent change = -32.4, 95% CI 2-sided [-45.3 to -16.4] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All-cause mortality and Adverse Event data collection is up to 11 weeks
Description: Analysis population consisted of all randomized participants who received at least 1 dose of study drug
Groups:
- Placebo: Matching Placebo for BLU-5937 administered orally BID for 4 days
Arm/Group | BLU-5937 - 25 mg | BLU-5937 - 50 mg | BLU-5937 - 100 mg | BLU-5937 - 200 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/61 | 0/60 | 0/58 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 0/60 | 0/58 | 1/61
Other Adverse Events (participants affected / at risk) | 10/61 | 14/61 | 15/60 | 10/58 | 19/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLU-5937 - 25 mg (N=61) | BLU-5937 - 50 mg (N=61) | BLU-5937 - 100 mg (N=60) | BLU-5937 - 200 mg (N=58) | Placebo (N=61)
colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | NA | NA | 1 (1) — colorectal cancer considered as not related to study drug was reported approximately 6 months after the last dose of study medication.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BLU-5937 - 25 mg (N=61) | BLU-5937 - 50 mg (N=61) | BLU-5937 - 100 mg (N=60) | BLU-5937 - 200 mg (N=58) | Placebo (N=61)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 4 (4) | 3 (3) | 7 (7)
Dysgeusia (Nervous system disorders) | 3 (3) | 5 (5) | 5 (5) | 4 (4) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4) | 3 (3) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 4 (4) | 4 (4) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No data collected as part of this study will be utilized in any written work, including publications, without the written consent of sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT03979638/Prot_SAP_000.pdf